CLINICAL TRIAL: NCT05282368
Title: Preparing Heart and Mind™: A Patient Engagement Pathway for Parents and Their Caregiving Partners After a Major Fetal Anomaly Diagnosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SON-2019-27260
Record Dates: First submitted 2022-02-07; First posted 2022-03-16 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Parent Mental Health
Keywords: parent; fetal anomaly; prenatal diagnosis; infant; heart disease; ehealth; intervention
MeSH Terms: conditions — Congenital Abnormalities; Heart Diseases

STUDY DESIGN:
Intervention Model Description: This small pilot study is designed as a mixed methods randomized controlled trial to estimate and test the effect of a nurse-guided PHM™ intervention on psychological distress and perceived caregiving competencies using longitudinal, repeated measures. Qualitative and quantitative data are expected to provide crucial insights regarding app usage patterns, interactions with the nurse interventionist, and impacts of the intervention on the individual/dyad.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (PHM) (Experimental): This pathway is intended to be a tool to enhance support for a mother/birthing person and her caregiving partner, facilitate communication with healthcare providers, and promote development of caregiving to optimize maternal-fetal, infant, and family health.
  Interventions: Behavioral: PHM™ Pathway
- Usual Care Group (UC) (No Intervention): The control group participants will receive care as usual.

INTERVENTIONS:
Behavioral: PHM™ Pathway — The technological platform referred to as Preparing Heart and Mind™ (PHM™) is designed as a patient engagement pathway. This platform includes GetWellNetwork's proprietary workflow engine, Patient Pathways™ and functionality of the Health Loop platform. Specifically, PHM™ will be created on a customized GetWellNetwork patient engagement pathway, getwell | Loop, which is a secure platform with a parent-facing app and an interactive dashboard for healthcare providers. The PHM™ getwell | Loop is a care program with chapters that incorporate interactive resources for patient information and education, trackers as touch points for psycho-social/educational support, and tailors care with condition-specific content, as well as action items.
  Arms: Intervention (PHM)

SUMMARY:
The purpose of this study is to test and evaluate the Preparing Heart and Mind™ (PHM™) patient engagement pathway as a nurse-guided intervention to lower psychological distress and enhance caregiving competencies among mothers/birthing persons and their caregiving partners after a major fetal anomaly diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* A study participant can include a pregnant person past 20 weeks of pregnancy (this includes a vulnerable population)
* Willing and able to comply with study procedures.
* Participants must be ≥ 18 years old.
* Participants must be able to read, write and speak English.
* Participants must have access, and ability to use a smartphone, tablet, or computer in a private location.
* The pregnant woman/person and her caregiving partner are planning for infant delivery and care.
* The fetal diagnosis of the major anomaly affects the heart (i.e., CCHD). See definition of CCHD included earlier in the protocol. Other anomalies could be present and potentially impair other organs.
* The infant's anomaly will likely require surgical and/or medical intervention within the first year of life.
* The fetus/infant is expected to live with surgical and/or medical intervention (this includes a vulnerable population).
* There may be genetic and/or chromosomal conditions in addition to the heart/structural anomalies

Exclusion Criteria:

* Pregnancy termination
* The fetal anomaly diagnosis is highly likely to result in fetal or infant demise shortly after birth.
* Adults lacking the capacity to consent
* Adults who do not have access to a smart phone, tablet, or device.
* Caregiving partner cannot enroll if mother is not enrolled

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Change in State-Trait Anxiety Inventory score | 12 weeks after birth
  State subscale, 20 items, 4-point scale; State Anxiety cut point score ≥40
Change in Center for Epidemiology Scale-Depression (CES-D) score | 12 weeks after birth
  20 items, 4-point scale; cut point score ≥16
Change in Impact of Event Scale score | 12 weeks after birth
  22 items, 4-point scale; cut point score ≥ 24

CONTACTS AND LOCATIONS:
Overall Officials: Anne C McKechnie, PhD, RN, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States